CLINICAL TRIAL: NCT03898193
Title: Single-Dose Open-label Randomized Crossover, in Two Periods and in Two Sequences, Single-Center Comparative Bioequivalence Study of Montelukast, 5 mg Chewable Tablets (Pharmtechnology LLC, Republic of Belarus), and Singulair®, 5 mg Chewable Tablets (Merck Sharp & Dohme B.V., the Netherlands), in Healthy Volunteers Under Fasting Conditions
Brief Title: Bioequivalence Study of Montelukast, 5 mg Chewable Tablets (Pharmtechnology LLC, Belarus), and Singulair®, 5 mg Chewable Tablets (Merck Sharp & Dohme B.V., the Netherlands), in Healthy Volunteers Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmtechnology LLC (Industry)
Collaborators: ClinPharmInvest, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: FRM-07-MONT v.2.1 01/29/2019
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-03

CONDITIONS: Healthy Adults
Keywords: Bioequivalence; Montelukast; Singulair
MeSH Terms: interventions — montelukast

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The participants and the investigator will not be blinded towards the identity of the study products. However, bioanalytical laboratory will be blinded towards identity of the study products administered.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence Test-Reference (TR) (Other): 17 participants (total number of enrolled volunteers - 34) assigned to sequence TR will receive a single 5 mg dose of the test product Montelukast (1 x 5 mg tablet) marked as T in period 1 and a single 5 mg dose of the reference product Singulair (1 x 5 mg tablet) marked as R in period 2. These treatments will be administered orally with 200 ml of water at ambient temperature, in the morning, following a 10-hour overnight fast. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Montelukast; Drug: Singulair
- Sequence Reference-Test (RT) (Other): 17 participants (total number of enrolled volunteers - 34) assigned to sequence RT will receive a single 5 mg dose of the reference product Singulair (1 x 5 mg tablet) marked as R in period 1 and a single 5 mg dose of the test product Montelukast (1 x 5 mg tablet) marked as T in period 2. These treatments will be administered orally with 200 ml of water at ambient temperature, in the morning, following a 10-hour overnight fast. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Montelukast; Drug: Singulair

INTERVENTIONS:
Drug: Montelukast — Montelukast, 5 mg Chewable Tablets, manufactured by Pharmtechnology LLC, Republic of Belarus
  Other Names: The test product
Drug: Singulair — Singulair, 5 mg Chewable Tablets, marketed by Merck Sharp & Dohme B.V., the Netherlands
  Other Names: The reference product

SUMMARY:
This is an open-label, randomized, single-center, single-dose, crossover, in two periods and in two sequences comparative study, where each participant is randomly assigned to the reference or the test formulation in each period of the study (sequences Test-Reference (TR) or Reference-Test (RT)), in order to evaluate if both formulations are bioequivalent.

DETAILED DESCRIPTION:
The objective of this study is to establish if two formulations of montelukast are bioequivalent. Also monitoring, registration and evaluation of adverse events will be performed.

The test formulation is Montelukast, 5 mg сhewable tablets (Pharmtechnology LLC, Belarus). The reference formulation is Singulair®, 5 mg сhewable tablets (Merck Sharp & Dohme B.V., the Netherlands). 34 healthy adult volunteers of both genders, with age ranging from 18 to 45 years old, will be divided into two cohorts with equal number of participants (17). Each participant in a cohort will receive single tablet (5 mg of montelukast) of the test or the reference product with 200 ml of water after an overnight fast of at least 10 hours, according to the pre-defined randomization list, i. e. 17 participants in each cohort will receive the test product and 17 participants in each cohort will receive the reference product in each of two periods of the study. Participants will fast 4 hours after administration of the study drugs during each study period. Standardized meals will be provided in each study period. Water will not be accessible to the participants 1 hour prior to administration of the study drugs and 2 hours after administration of the study drugs in each period. In each period blood samples will be collected withing 30 minutes before dosing and 0.5, 1.00, 1.5, 1.75, 2.00, 2.25, 2.5, 2.75, 3.00, 3.25, 3.5, 4.00, 4.5, 5.00, 6.00, 8.00, 12.00, 16.00, 24.00 hours after dosing (total number: 20). The washout period will be 7 days.

At the bio-analytical stage, a validated High Performance Liquid Chromatography with Tandem Mass Spectrometry detection (HPLC/MS) method will be used to determine plasma concentrations of montelukast. At all stages of working with biological samples measures to protect montelukast from daylight exposure should be provided.

ANOVA will be performed on log transformed pharmacokinetic parameters Cmax, Area Under the pharmacokinetic Curve from the beginning of the study to the time of the last measured concentration (AUC0-t) and 90% confidence interval will be constructed for the ratio of geometric means of the test and the reference products, obtained from the log-transformed data. Bioequivalence will be concluded if the ratio estimate as well as its 90% confidence interval for montelukast falls within the acceptable range of 80.00% to 125.00% for Cmax and AUC0-t

ELIGIBILITY:
Inclusion Criteria:

* Healthy caucasian men or women aged between 18 to 45 years
* Subjects having no clinically significant medical history and no clinically significant abnormalities in general physical examination, laboratory assessments and imaging studies
* Body mass index 18.5-30 kg/m² with body mass >45 kg and ≤100 kg
* Non-breastfeeding women
* Non-pregnant women (negative pregnancy test)
* If subject is a female and is of childbearing potential, she should practice an acceptable non-hormonal method of birth control for the duration of the study (the entire time from the moment of signing the informed consent form and within 14 days after the completion of the study), such as a combination of male condom and diaphragm with spermicide, the use of which has begun at least 30 days before the start of participation in the study
* If subject is a male and has a female partner of childbearing potential, he should be practicing an acceptable method of birth control for the duration of the study (the entire time from the moment of signing the informed consent form and within 14 days after the completion of the study), such as a double barrier method of birth control or sexual continence during the whole study and within 14 days after completion of the study
* Subjects are able to understand the requirements of the study, to sign a written informed consent, and also to accept all the restrictions imposed during the course of the study, and to agree to return for the required investigations

Exclusion Criteria:

* Subjects with a known history of allergic disorders
* Hypersensitivity to montelukast or to any of the excipients of the test and the reference product
* Subjects with a known history of drug intolerance
* Dehydration due to diarrhea, vomiting, or another cause in the last 24 hours before the beginning of the first period of the study
* Subjects with history of psychiatric disorders
* History of convulsions, epilepsy and any other neurological disorders
* Adherence to any low sodium diet for 2 weeks before starting research, or adherence to a special diet (for example, vegetarian, vegan, with restriction of the use of salt) or lifestyle (work at night, extreme physical exertion)
* Use of gestagen-containing injectable hormonal contraceptives, implants, intrauterine hormonal therapeutic systems within 6 months prior to start of the study
* Female subjects of childbearing potential having unprotected intercourse with an unsterilized male partner within 30 days prior to start of the study
* Consumption of xanthine-containing foods and drinks (tea, coffee, coca-cola, chocolate) within 72 hours prior to start of the first period of the study
* Consumption of citrus fruits (including grapefruit and grapefruit juice) and cranberries (including cranberry juice and other cranberry drinks) within 14 days prior to start of the study
* Acute and chronic cardiovascular, respiratory, gastrointestinal diseases, neuroendocrine disorders, renal and/or hepatic impairment, blood system disorders
* Other conditions which, according to the researcher's judgment, may affect absorption, distribution, biotransformation and elimination of any formulation or increase risks of deterioration of volunteer's condition
* Surgical interventions on the gastrointestinal tract with the exception of appendectomy
* Acute infectious diseases less than 4 weeks prior to the start of the study
* ECG abnormalities
* Sitting systolic blood pressure < 100 mm Hg or > 130 mm Hg and/or sitting diastolic blood pressure < 70 mm Hg or > 90 mm Hg
* Heart rate <60 or >80 beats per minute at screening check-in
* Use of liver enzyme inducers and inhibitors, in particular isoenzyme CYP3A4 (inducers: omeprazole, cimetidine, products containing the extract of Hypericum perforatum, barbiturates, carbamazepine, phenytoin, glucocorticoids; inhibitors: antiviral drugs, clarithromycin, ciprofloxacin, gestodene etc.) within 2 months prior to the start of the study
* Use of any systemic drugs within 14 days prior to the start of the study
* Use of Over-The-Counter (OTC) drugs, including herbs and nutritional supplements within 7 days prior to the First Dosing Date (including vitamins and natural food additives, phyto supplements,herbal preparations such as, cat's claw, angelica officinalis, oenothera, feverfew, garlic, ginger, ginkgo, red clover, horse chestnut, green tea, ginseng)
* Donation of plasma or blood (450 ml or more) within 2 months prior to the start of the study
* Intake of more than 10 units alcohol per week (1 unit of alcohol is equivalent to ½ liter of beer, 200 ml dry wine or 50 ml of spirits) or history of alcoholism, drug addiction, drug abuse
* Intake of more than 10 units alcohol per week (1 unit of alcohol is equivalent to ½ liter of beer, 200 ml dry wine or 50 ml of spirits) or history of alcoholism, drug addiction, drug abuse
* Smoking more than 10 cigarettes per day
* Participation in other clinical trials of medicines within 3 months prior to the start of the study
* Positive test for syphilis, hepatitis B, hepatitis C or HIV
* Positive pregnancy test (for female subjects with childbearing potential)
* Breast-feeding
* In the case of using of oral hormonal contraceptives, they should be withdrawn 2 months prior to the start of the study
* Positive test for alcohol in exhaled air
* Positive urinary screen test for the content of narcotic and potent substances during screening and at each arrival at the research stage
* The values of standard laboratory and instrumental parameters that go beyond the reference values of the local clinical laboratory for laboratory parameters and the conventional reference values for instrumental parameters
* History of phenylketonuria

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-03-23 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
Cmax of montelukast for the test and the reference products | Time points: 0.00 (withing 30 minutes before dosing) and 0.5, 1.00, 1.5, 1.75, 2.00, 2.25, 2.5, 2.75, 3.00, 3.25, 3.5, 4.00, 4.5, 5.00, 6.00, 8.00, 12.00, 16.00, 24.00 hours after dosing
  Maximum concentration in plasma among observed concentrations at pre-specified time points
AUC0-t of montelukast for the test and the reference products | Time points: 0.00 (withing 30 minutes before dosing) and 0.5, 1.00, 1.5, 1.75, 2.00, 2.25, 2.5, 2.75, 3.00, 3.25, 3.5, 4.00, 4.5, 5.00, 6.00, 8.00, 12.00, 16.00, 24.00 hours after dosing
  Area under the plasma concentration versus time curve from time 0 to the last measured concentration

SECONDARY OUTCOMES:
AUC0-∞ of montelukast for the test and the reference products | Time points: 0.00 (withing 30 minutes before dosing) and 0.5, 1.00, 1.5, 1.75, 2.00, 2.25, 2.5, 2.75, 3.00, 3.25, 3.5, 4.00, 4.5, 5.00, 6.00, 8.00, 12.00, 16.00, 24.00 hours after dosing
  Area under the plasma concentration versus time curve from time 0 to infinite time
Tmax of montelukast for the test and the reference products | Time points: 0.00 (withing 30 minutes before dosing) and 0.5, 1.00, 1.5, 1.75, 2.00, 2.25, 2.5, 2.75, 3.00, 3.25, 3.5, 4.00, 4.5, 5.00, 6.00, 8.00, 12.00, 16.00, 24.00 hours after dosing
  Time to maximum measured plasma concentration
T1/2 of montelukast for the test and the reference products | Time points: 0.00 (withing 30 minutes before dosing) and 0.5, 1.00, 1.5, 1.75, 2.00, 2.25, 2.5, 2.75, 3.00, 3.25, 3.5, 4.00, 4.5, 5.00, 6.00, 8.00, 12.00, 16.00, 24.00 hours after dosing
  Elimination or terminal half-life
Kel of montelukast for the test and the reference products | Time points: 0.00 (withing 30 minutes before dosing) and 0.5, 1.00, 1.5, 1.75, 2.00, 2.25, 2.5, 2.75, 3.00, 3.25, 3.5, 4.00, 4.5, 5.00, 6.00, 8.00, 12.00, 16.00, 24.00 hours after dosing
  Elimination rate constant
AUCresid of montelukast for the test and the reference products | Time points: 0.00 (withing 30 minutes before dosing) and 0.5, 1.00, 1.5, 1.75, 2.00, 2.25, 2.5, 2.75, 3.00, 3.25, 3.5, 4.00, 4.5, 5.00, 6.00, 8.00, 12.00, 16.00, 24.00 hours after dosing
  Residual area under the pharmacokinetic curve from the time of the last measured concentration to infinite time
Number of treatment-related adverse events (AE) for the test and the reference products as assessed by guidance predefined in the protocol | 8 days
  An AE is defined as any untoward medical occurrence in a subject will be administered an investigational product and which does not necessarily have a causal relationship with the treatment. The data from subjects who will take at least one investigational product will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Khokhlov, Principal Investigator — ClinPharmInvest, LLC
Locations (1):
- State Autonomous Healthcare Facility of the Yaroslavl Region "Clinical Hospital No. 2", Yaroslavl, Yaroslavl Oblast, Russia